CLINICAL TRIAL: NCT07360119
Title: Total Pancreatectomy With Islet Autotransplantation (TPIAT) for Patients With Periampullary Neoplasms at High Risk for Pancreaticojejunostomy Leakage After Pancreaticoduodenectomy: a Single-center, Prospective, Single-Arm, Observational Study
Brief Title: Total Pancreatectomy With Islet Autotransplantation (TPIAT) for High-Risk Patients With Pancreatic Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00543437
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Periampullary Neoplasms; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TPIAT for Patients with High-Risk Periampullary Neoplasms (Experimental): This single-arm study investigates the outcomes of Total Pancreatectomy with Islet Autotransplantation (TPIAT) in patients diagnosed with high-risk periampullary neoplasms. The intervention aims to eliminate the risk of postoperative pancreatic fistula and preserve endocrine function, while assessing safety and feasibility. Participants will undergo TPIAT via either open or robotic surgical techniques, and various postoperative metrics will be evaluated over a 12-month period.
  Interventions: Procedure: Total Pancreatectomy with Islet Autotransplantation (TPIAT)

INTERVENTIONS:
Procedure: Total Pancreatectomy with Islet Autotransplantation (TPIAT) — This intervention involves a total pancreatectomy with subsequent islet autotransplantation for patients diagnosed with high-risk periampullary neoplasms. The procedure is performed following strict surgical protocols and includes resection of the pancreas while aiming to eliminate the risk of postoperative pancreatic fistula (POPF). Islet cells are isolated from the nontumorous pancreatic tissue and infused into the portal vein to maintain endocrine function, thus reducing the likelihood of brittle diabetes post-surgery. Patient outcomes will be evaluated for safety, metabolic control, and overall quality of life over a 12-month follow-up period.

SUMMARY:
This is a single-center, prospective, single-arm study evaluating the safety and feasibility of total pancreatectomy with islet autotransplantation (TPIAT) in carefully selected adult patients with periampullary neoplasms who are considered at high risk for postoperative pancreatic fistula after pancreaticoduodenectomy. Eligible patients will undergo open or robotic TPIAT as part of the patient's surgical management. Perioperative outcomes, postoperative complications, metabolic outcomes, and early oncologic outcomes will be collected prospectively as part of routine clinical care and analyzed to assess the safety and feasibility of this approach.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older.
* Patients with periampullary neoplasms requiring pancreaticoduodenectomy, including but not limited to:
* Distal bile duct adenocarcinoma
* Duodenal adenocarcinoma
* Leiomyosarcoma of the duodenum
* Pancreatic neuroendocrine neoplasms
* Ampullary adenoma
* Duodenal gastrointestinal stromal tumor (GIST)
* High-risk Intraductal Papillary Mucinous Neoplasm (IPMN) as per Fukuoka criteria
* Mucinous cystic neoplasm
* Serous cystadenoma
* Presence of soft pancreatic tissue and a main pancreatic duct ≤ 2 mm based on preoperative imaging.
* Adequate islet function with measurable C-peptide preoperatively to justify islet isolation and transplant.

Exclusion Criteria:

* Pregnancy
* Active alcohol or illicit drug use
* Poorly controlled psychiatric illness that limits compliance with care
* Pre-existing insulin-dependent diabetes with absent C-peptide
* Portal vein thrombosis or significant portal hypertension
* Contraindications to major surgery
* Body Mass Index (BMI) > 35 kg/m².

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2031-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Complications | Within 90 days post-surgery.
  The incidence of postoperative complications within 90 days following Total Pancreatectomy with Islet Autotransplantation (TPIAT) will be assessed. Complications will be defined and graded according to the Clavien-Dindo classification system. The goal is to evaluate the safety and feasibility of TPIAT in high-risk patients with periampullary neoplasms.

SECONDARY OUTCOMES:
Length of Hospital Stay | Within 90 days post-surgery.
  This measure will track the total number of days patients remain hospitalized following TPIAT. The data will help evaluate the procedure's impact on recovery time.

CONTACTS AND LOCATIONS:
Overall Officials: Jin He, MD, Principal Investigator — SKCCC Johns Hopkins Medical Institution